CLINICAL TRIAL: NCT05538663
Title: A Randomized Phase III Trial of Intravesical BCG veRsus Intravesical Docetaxel and GEmcitabine Treatment in BCG Naïve High Grade Non-Muscle Invasive Bladder Cancer (BRIDGE)
Brief Title: Intravesical BCG vs GEMDOCE in NMIBC
Acronym: BRIDGE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA8212; U10CA180820 (NIH); NCI-2022-04864 (Other: NCI)
Record Dates: First submitted 2022-08-25; First posted 2022-09-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Non-muscle-invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine; Docetaxel; BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Gemcitabine + Docetaxel
  Interventions: Drug: Gemcitabine; Drug: Docetaxel
- Arm B (Experimental): BCG
  Interventions: Drug: Bacillus Calmette Guerin

INTERVENTIONS:
Drug: Gemcitabine — Intravesical once a week for 6 consecutive weeks followed by monthly instillations during maintenance for 2 years
  Other Names: GEMZAR
  Arms: Arm A
Drug: Docetaxel — Intravesical once a week for 6 consecutive weeks followed by monthly instillations during maintenance for 2 years
  Other Names: Taxotere
  Arms: Arm A
Drug: Bacillus Calmette Guerin — intravesical once a week for 6 consecutive weeks during induction followed by weekly instillations for 3 consecutive weeks at months 3, 6, 12, 18, 24, 30, and 36 months
  Other Names: BCG
  Arms: Arm B

SUMMARY:
The study hypothesis is that BCG naïve non-muscle invasive bladder cancer (NMIBC) patients treated with intravesical Gemcitabine + Docetaxel (GEMDOCE) will result in a non-inferior event-free survival (EFS) compared to standard treatment with intravesical BCG. The purpose of this study is to test whether Gemcitabine + Docetaxel is a better or worse treatment than the usual BCG therapy approach. The primary objective of this study is to determine the event free survival (EFS) of BCG-naïve high grade non-muscle invasive bladder cancer patients treated with intravesical BCG vs Gemcitabine + Docetaxel. Secondary objectives are as follows: to compare changes in cancer-specific and bladder cancer-specific QOL from baseline to treatment between BCG-naïve high grade NMIBC patients receiving BCG and GEMDOCE, to determine the cystectomy free survival (CFS) of BCG-naïve high grade NMIBC patients treated with intravesical BCG vs GEMDOCE, to determine the progression free survival (PFS) of BCG-naïve high grade NMIBC patients treated with intravesical BCG vs GEMDOCE, and to determine the safety and toxicity of BCG-naïve high grade NMIBC patients treated with intravesical BCG vs GEMDOCE.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the event free survival (EFS) of BCG-naïve high grade non-muscle invasive bladder cancer patients treated with intravesical BCG vs Gemcitabine + Docetaxel. Secondary objectives are as follows: to compare changes in cancer-specific and bladder cancer-specific QOL from baseline to treatment between BCG-naïve high grade NMIBC patients receiving BCG and GEMDOCE, to determine the cystectomy free survival (CFS) of BCG-naïve high grade NMIBC patients treated with intravesical BCG vs GEMDOCE, to determine the progression free survival (PFS) of BCG-naïve high grade NMIBC patients treated with intravesical BCG vs GEMDOCE, and to determine the safety and toxicity of BCG-naïve high grade NMIBC patients treated with intravesical BCG vs GEMDOCE

ELIGIBILITY:
Inclusion Criteria:

* Patient must be > 18 years of age.
* Patient must have histologically confirmed high-grade non-muscle invasive urothelial carcinoma of the bladder (HgTa, HGT1, CIS, HgTa + CIS, or HGT1 + CIS stage) on transurethral resection of bladder tumor (TURBT) obtained within 90 days prior to randomization.
* Patient must have all visible papillary tumor resected by the treating urologist at the site registering the patient to this protocol prior to randomization. If the treating urologist did not perform the TURBT as outlined in Section 3.1.3, the treating urologist must perform a cystoscopy within 28 days prior to randomization to confirm the absence of visible papillary disease.
* Patient must have not received prior intravesical therapy for bladder cancer, with the exception of perioperative chemotherapy at the time of TURBT.
* Patients with high grade T1 disease must have undergone a restaging TURBT within 90 days prior to Step 1 randomization.

NOTE: Patients with high grade T1 disease who undergo a restaging TURBT that shows no residual cancer in the restaging TURBT specimen are eligible.

* Patient must not have pure squamous cell carcinoma or adenocarcinoma.
* Patient must not have any component of neuroendocrine carcinoma (i.e., small cell or large cell).
* Patient must not have any component of sarcomatoid, micropapillary, or plasmacytoid variant histology.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patient must have ECOG Performance Status 0-2.
* Patient may have received prior systemic gemcitabine or docetaxel use if it was for a non-bladder malignancy.
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
* Patient must have adequate organ and marrow function as defined below (these labs must be obtained ≤ 28 days prior to randomization):

Leukocytes ≥ 3,000/mcL Leukocytes:__________ Date of Test:__________ Absolute neutrophil count (ANC) ≥ 1,500/mcL ANC:__________ Date of Test:__________ Platelets ≥ 70,000/mcL Platelets:__________ Date of Test:__________ Total Bilirubin ≤ institutional upper limit of normal (ULN) Total Bilirubin:__________ Institutional ULN:_________ Date of Test:__________ AST(SGOT)/ALT(SGPT) ≤ 3.0 × institutional ULN AST:_______ Institutional ULN:_________ Date of Test:_______ ALT: _______Institutional ULN:_________

* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

Exclusion Criteria:

* Patient must not have any prior or current history of muscle-invasive (i.e., T2, T3, T4), locally advanced unresectable, or metastatic urothelial carcinoma as assessed on radiographic imaging obtained within 90 days prior to randomization. The radiographic imaging includes a CT Scan OR MRI of the abdomen/pelvis with intravenous contrast.

NOTE: If a patient's renal function does not permit the administration of intravenous contrast, either a CT scan or MRI of the abdomen/pelvis without intravenous contrast is acceptable.

NOTE: Patients with a history of non-invasive (Ta, Tis) upper tract urothelial carcinoma that has been definitively treated with at least one post-treatment disease assessment (i.e., either cytology, biopsy, or imaging) that demonstrates no evidence of residual disease are eligible.

- Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy.

A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Patient of child bearing potential? ______ (Yes or No) Date of blood test or urine study: ___________

* Patient must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study. In addition,patients on Arm A must continue contraception measures for six months after the last dose of GEMDOCE for patients of child-bearing potential and continue for three month after the last dose of GEMDOC for male patients with partners of child-bearing potential. All patients must not breastfeed during their time on protocol treatment.
* Patient must not have a history of severe hypersensitivity reactions to docetaxel or drugs formulated with polysorbate 80.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival | 2 years
  To determine the event free survival (EFS) of BCG-naïve high grade non-muscle invasive bladder cancer (NMIBC) patients treated with intravesical BCG vs GEMDOCE.

SECONDARY OUTCOMES:
Quality of Life FACT-G | 3 years
  To compare changes in cancer-specific QOL from baseline to treatment between BCG-naïve high grade NMIBC patients receiving BCG and GEMDOCE.
Cystectomy free survival | 3 years
  To determine the cystectomy free survival (CFS) of BCG-naïve high grade NMIBC patients treated with intravesical BCG vs GEMDOCE.
Progression Free Survival | 3 years
  To determine the progression free survival (PFS) of BCG-naïve high grade NMIBC patients treated with intravesical BCG vs GEMDOCE
Quality of Life EORTC NMIBC-24 | 3 years
  To compare changes in bladder cancer-specific QOL from baseline to treatment between BCG-naïve high grade NMIBC patients receiving BCG and GEMDOCE.

CONTACTS AND LOCATIONS:
Locations (229):
- United States (229):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Mercy Cancer Center, Merced, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Mercy Health - Paducah Cancer Center, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Ochsner LSU Health - Cancer Treatment Center, Shreveport, Louisiana
  - Maine Medical Partners Urology, South Portland, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center-Rockledge, Rockledge, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC Health Florence Medical Center, Florence, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - MD Anderson in The Woodlands, Conroe, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Jefferson Healthcare, Port Townsend, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koti M, Robert Siemens D. A Step Closer to Predicting Progression After Bacillus Calmette-Guerin Immunotherapy in High-risk Non-muscle-invasive Bladder Cancer. Eur Urol. 2023 Nov;84(5):447-448. doi: 10.1016/j.eururo.2023.06.017. Epub 2023 Jul 1. PMID 37400353